CLINICAL TRIAL: NCT06228807
Title: Exploring Clinical Characteristics and Predictors of Adverse Outcomes in Patients Diagnosed With Heart Failure With Preserve Ejection Fraction (HFpEF)
Brief Title: Clinical Characteristics and Predictors of Adverse Outcomes in HFpEF
Status: Completed | Type: Observational
Sponsor: Ya-Wei Xu (Other)
Responsible Party: Sponsor-Investigator, Ya-Wei Xu, Chief Physician, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Other Study IDs: HFpEF-CCPO
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: risk predictors; mortality
MeSH Terms: interventions — Health Records, Personal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HFpEF patients with metabolic abnormalities
  Interventions: Combination Product: The study involved a comparison of clinical characteristics, medical history, laboratory biomarkers, echocardiographic measurements, angiographic findings, and clinical outcomes between two groups.
- HFpEF patients without metabolic abnormalities
  Interventions: Combination Product: The study involved a comparison of clinical characteristics, medical history, laboratory biomarkers, echocardiographic measurements, angiographic findings, and clinical outcomes between two groups.

INTERVENTIONS:
Combination Product: The study involved a comparison of clinical characteristics, medical history, laboratory biomarkers, echocardiographic measurements, angiographic findings, and clinical outcomes between two groups. — Differences in clinical characteristics, history, laboratory biomarkers, echocardiographic measurements, angiographic findings, coronary microvascular function using caIMR and clinical outcomes were assessed between the two groups to identify potential risk factors. Subsequently, the incidence of clinical outcomes and mortality was compared. Univariate logistic regression and multivariate logistic regression analyses, adjusted for significant risk factors, were conducted to identify independent predictive factors. Finally, a Receiver Operating Characteristic (ROC) curve was generated, and the area under the curve was evaluated to assess the predictive accuracy of the regression model.

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) is a prevalent form of heart failure characterized by impaired left ventricle pressures and diastolic dysfunction. Despite its increasing prevalence, effective treatment options for HFpEF remain limited, probably due to its heterogenous underlying pathological etiology involving chronic systemic inflammation and metabolic dysregulation. Identifying new predictors of poor prognosis is crucial for risk stratification and tailored management.

DETAILED DESCRIPTION:
The prognosis for HFpEF is concerning, marked by significant mortality and frequent hospital readmissions. The exact mechanisms underlying HFpEF remain unresolved. The clinical syndrome arises from intricate interactions among various risk factors, leading to organ dysfunction and clinical symptoms. Common co-morbidities, including atrial fibrillation, diabetes, chronic kidney disease, and obesity, may influence HFpEF pathophysiology. Recent discussions suggest an inflammatory-metabolic phenotype in HFpEF, characterized by heightened inflammatory biomarkers, insulin resistance, hyperglycemia, hyperlipidemia, microvascular endothelial and vascular dysfunction, atherosclerosis, consequently leading to significant myocardial damage. However, there is still a lack of clinical risk predictors associated with metabolic phenotype within HFpEF.

The aim of this study is to investigate the impact of parameters reflecting the metabolic phenotype, coronary microvascular dysfunction in HFpEF and establish their correlation with clinical outcomes. The objective is to identify novel predictors for adverse prognosis in HFpEF, potentially serving as targets for drug therapy. This research aims to pave the way for targeted drug interventions in cardiometabolic diseases, offering new avenues for therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with HFpEF; Diagnostic criteria for HFpEF

  * Presence of heart failure signs/symptoms symptoms
  * Preserved left ventricular ejection fraction (EF) ≥50%
  * BNP≥35 pg/mL and/or NTproBNP≥125 pg/mL;
  * At least one additional criteria: presence of cardiac functional and structural abnormalities or diastolic dysfunction.

Exclusion Criteria:

* LVEF lower than 50%
* Patients with serious hepatic and renal failure,
* Non-cardiac causes of dyspnea, such as, asthma
* Primary pulmonary hypertension.
* Severe valvular heart disease.
* Pericardial disease.
* Recent history of myocardial infarction.
* Coronary artery disease (stenosis>50).
* Reduced contrast opacification (for caIMR assessment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Heart failure with preserved ejection fraction(HFpEF)
Sampling Method: Non-Probability Sample
Enrollment: 584 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Composite Events | From the time of hospital discharge until the event of specific outcome, death, or loss to follow up, maximum 10 years.
  The composite events include a composite of all-cause mortality (death due to any cause), cardiovascular mortality (death due to cardiac cause), and heart failure rehospitalization.

IPD SHARING:
Plan to Share IPD: No